CLINICAL TRIAL: NCT01939704
Title: Community to Clinic Linkage Program at SFGH
Acronym: CCLiP@SFGH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 13-11628
Record Dates: First submitted 2013-09-06; First posted 2013-09-11 (Estimated); Last update posted 2019-12-18 (Actual); Status verified 2019-12

CONDITIONS: Family's Connection to Community Resources and Public Benefits; Caregiver Satisfaction and Connectedness to Clinic; Child Health Care Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Pediatric Primary Care Control (No Intervention): Baseline survey with a social needs assessment, health care status, health care satisfaction and health care utilization assessment and two telephone-based follow up surveys at 3 and 6 months.
- Pediatric Urgent Care Control (No Intervention): Baseline survey with a social needs assessment, health care status, health care satisfaction and health care utilization assessment and two telephone-based follow up surveys at 3 and 6 months.
- Pediatric Primary Care Intervention (Experimental): Baseline survey that includes social needs assessment, health care status, health care satisfaction and health care utilization assessment; 30 minute on-site intervention, twice monthly follow-up phone calls for up to 3 months to help address social needs
  Interventions: Other: Pediatric Primary Care Intervention
- Pediatric Urgent Care Intervention (Experimental): Baseline survey that includes social needs assessment, health care status, health care satisfaction and health care utilization assessment; 30 minute on-site intervention, twice monthly follow-up phone calls for up to 3 months to help address social needs
  Interventions: Other: Pediatric Urgent Care Intervention

INTERVENTIONS:
Other: Pediatric Primary Care Intervention — 30 minute on-site intervention with biweekly follow up phone calls to address social needs and health care status.
  Arms: Pediatric Primary Care Intervention
Other: Pediatric Urgent Care Intervention — 3 months of intervention protocol, including a 30 minute on-site intervention and twice monthly phone calls to address social needs and health care status.
  Arms: Pediatric Urgent Care Intervention

SUMMARY:
It is increasingly clear that the environment in which a child lives, plays, and goes to school has a significant impact on their health. With the implementation of a Community to Clinic Linkage Program (CCLiP) in the SFGH Pediatrics Clinics, we will routinely address Social Determinants of Health when families present. We will randomize patients to receive either the CCLiP intervention or standard of care. We will evaluate programmatic outcome, health care utilization data and return on investment data. We hypothesize that by addressing the environmental and social factors that contribute to health within the setting of the medical home, we will be able to better connect families to community resources, enable more appropriate use of healthcare resources, improve health status, and enhance patient satisfaction.

DETAILED DESCRIPTION:
We are proposing a 4-arm, 18 month randomized control clinical trial to address social determinants of health, improve health status and health care satisfaction, and change health care utilization patterns in the Pediatric Urgent Care and Primary Care Clinics at San Francisco General Hospital. We will compare our CCLiP protocol to standard of care in both the Pediatric Primary Care Clinic & Urgent Care. All arms (intervention and control) include a baseline survey including social needs assessment, health care status, health care satisfaction and health care utilization assessment; and two telephone-based follow up surveys at 3 and 6 months. Patients in the intervention arms (whether in urgent care or primary care) will receive a maximum of 3 months of intervention protocol which includes a 30 minute on-site intervention at time of enrollment in addition to twice monthly follow-up phone calls for up to 3 months to help address social needs. Patients in all arms will receive 3 and 6-month follow up surveys.

ELIGIBILITY:
Inclusion Criteria:

* English or Spanish Speaking
* Parent/caregiver accompanying an SFGH Primary Care or Urgent Care Clinic patient 0-17 years old
* Consenting adult over or equal to 18 years old

Exclusion Criteria:

* Non-English or non-Spanish speaking caregiver
* Caregiver under age 18
* Caregiver accompanying patient is not familiar with the child's living situation
* Family participated in study previously
* Non-San Francisco resident
* Foster child or child in clinic for a child protective clearance exam

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1809 (Actual)
Dates: Start 2013-10; Primary Completion 2015-09 (Actual); Study Completion 2019-10 (Actual)

PRIMARY OUTCOMES:
Family's connection to community resources and public benefits | up to 6 months post base-line
  This will be assessed at 3 months and 6 months post-enrollment by phone administered questionnaires.

SECONDARY OUTCOMES:
Child health care utilization | up to 6 months
  This will be assessed at 3 months and 6 months post-enrollment by phone administered questionnaires.
Child health status | up to 6 months
  This will be assessed at 3 months and 6 months post-enrollment by phone administered questionnaires.

OTHER OUTCOMES:
Caregiver satisfaction with care/connectedness to clinical setting | up to 6 months
  This will be assessed at 3 months and 6 months post-enrollment by phone administered questionnaires.

CONTACTS AND LOCATIONS:
Overall Officials: Laura M Gottlieb, MD, MPH, Principal Investigator — University of California, San Francisco
Locations (1):
- San Francisco General Hospital, San Francisco, California, United States

REFERENCES:
- [Background] Larson K, Russ SA, Crall JJ, Halfon N. Influence of multiple social risks on children's health. Pediatrics. 2008 Feb;121(2):337-44. doi: 10.1542/peds.2007-0447. PMID 18245425
- [Background] Wood PR, Smith LA, Romero D, Bradshaw P, Wise PH, Chavkin W. Relationships between welfare status, health insurance status, and health and medical care among children with asthma. Am J Public Health. 2002 Sep;92(9):1446-52. doi: 10.2105/ajph.92.9.1446. PMID 12197971
- [Background] Cook JT, Frank DA, Berkowitz C, Black MM, Casey PH, Cutts DB, Meyers AF, Zaldivar N, Skalicky A, Levenson S, Heeren T. Welfare reform and the health of young children: a sentinel survey in 6 US cities. Arch Pediatr Adolesc Med. 2002 Jul;156(7):678-84. doi: 10.1001/archpedi.156.7.678. PMID 12090835
- [Background] Frank DA, Neault NB, Skalicky A, Cook JT, Wilson JD, Levenson S, Meyers AF, Heeren T, Cutts DB, Casey PH, Black MM, Berkowitz C. Heat or eat: the Low Income Home Energy Assistance Program and nutritional and health risks among children less than 3 years of age. Pediatrics. 2006 Nov;118(5):e1293-302. doi: 10.1542/peds.2005-2943. PMID 17079530
- [Background] Meyers A, Cutts D, Frank DA, Levenson S, Skalicky A, Heeren T, Cook J, Berkowitz C, Black M, Casey P, Zaldivar N. Subsidized housing and children's nutritional status: data from a multisite surveillance study. Arch Pediatr Adolesc Med. 2005 Jun;159(6):551-6. doi: 10.1001/archpedi.159.6.551. PMID 15939854
- [Background] Garg A, Butz AM, Dworkin PH, Lewis RA, Serwint JR. Screening for basic social needs at a medical home for low-income children. Clin Pediatr (Phila). 2009 Jan;48(1):32-6. doi: 10.1177/0009922808320602. Epub 2008 Jun 19. PMID 18566347
- [Background] Lawton E, Leiter K, Todd J, Smith L. Welfare reform: advocacy and intervention in the health care setting. Public Health Rep. 1999 Nov-Dec;114(6):540-9. doi: 10.1093/phr/114.6.540. PMID 10670622
- [Background] Hanson M, Lawton E. Between a rock and a hard place: The prevalence and severity of unmet legal needs in the pediatric emergency department setting. Medical Legal Partnership for Children, 2007.
- [Background] Fleegler EW, Lieu TA, Wise PH, Muret-Wagstaff S. Families' health-related social problems and missed referral opportunities. Pediatrics. 2007 Jun;119(6):e1332-41. doi: 10.1542/peds.2006-1505. PMID 17545363
- [Background] Garg A, Butz AM, Dworkin PH, Lewis RA, Thompson RE, Serwint JR. Improving the management of family psychosocial problems at low-income children's well-child care visits: the WE CARE Project. Pediatrics. 2007 Sep;120(3):547-58. doi: 10.1542/peds.2007-0398. PMID 17766528
- [Background] Bikson K, McGuire J, Blue-Howells J, Seldin-Sommer L. Psychosocial problems in primary care: patient and provider perceptions. Soc Work Health Care. 2009;48(8):736-49. doi: 10.1080/00981380902929057. PMID 20182986
- [Background] Keller D, Jones N, Savageau JA, Cashman SB. Development of a brief questionnaire to identify families in need of legal advocacy to improve child health. Ambul Pediatr. 2008 Jul-Aug;8(4):266-9. doi: 10.1016/j.ambp.2008.04.004. Epub 2008 May 27. PMID 18644550
- [Background] Black MM, Cutts DB, Frank DA, Geppert J, Skalicky A, Levenson S, Casey PH, Berkowitz C, Zaldivar N, Cook JT, Meyers AF, Herren T; Children's Sentinel Nutritional Assessment Program Study Group. Special Supplemental Nutrition Program for Women, Infants, and Children participation and infants' growth and health: a multisite surveillance study. Pediatrics. 2004 Jul;114(1):169-76. doi: 10.1542/peds.114.1.169. PMID 15231924
- [Background] Jones SJ, Jahns L, Laraia BA, Haughton B. Lower risk of overweight in school-aged food insecure girls who participate in food assistance: results from the panel study of income dynamics child development supplement. Arch Pediatr Adolesc Med. 2003 Aug;157(8):780-4. doi: 10.1001/archpedi.157.8.780. PMID 12912784
- [Background] Cook JT, Frank DA, Berkowitz C, Black MM, Casey PH, Cutts DB, Meyers AF, Zaldivar N, Skalicky A, Levenson S, Heeren T, Nord M. Food insecurity is associated with adverse health outcomes among human infants and toddlers. J Nutr. 2004 Jun;134(6):1432-8. doi: 10.1093/jn/134.6.##. PMID 15173408
- [Background] Cook JT, Frank DA, Levenson SM, Neault NB, Heeren TC, Black MM, Berkowitz C, Casey PH, Meyers AF, Cutts DB, Chilton M. Child food insecurity increases risks posed by household food insecurity to young children's health. J Nutr. 2006 Apr;136(4):1073-6. doi: 10.1093/jn/136.4.1073. PMID 16549481
- [Derived] Pantell MS, Hessler D, Long D, Alqassari M, Schudel C, Laves E, Velazquez DE, Amaya A, Sweeney P, Burns A, Harrison FL, Adler NE, Gottlieb LM. Effects of In-Person Navigation to Address Family Social Needs on Child Health Care Utilization: A Randomized Clinical Trial. JAMA Netw Open. 2020 Jun 1;3(6):e206445. doi: 10.1001/jamanetworkopen.2020.6445. PMID 32478849
- [Derived] Gottlieb L, Hessler D, Long D, Laves E, Burns A, Amaya A, Schudel C, Sweeney P, Adler N. Are acute care settings amenable to addressing patient social needs: A sub-group analysis. Am J Emerg Med. 2018 Nov;36(11):2108-2109. doi: 10.1016/j.ajem.2018.03.034. Epub 2018 Mar 16. No abstract available. PMID 29576258
- [Derived] Gottlieb LM, Hessler D, Long D, Laves E, Burns AR, Amaya A, Sweeney P, Schudel C, Adler NE. Effects of Social Needs Screening and In-Person Service Navigation on Child Health: A Randomized Clinical Trial. JAMA Pediatr. 2016 Nov 7;170(11):e162521. doi: 10.1001/jamapediatrics.2016.2521. Epub 2016 Nov 7. PMID 27599265